CLINICAL TRIAL: NCT04506892
Title: Quantitation of Glymphatic Functioning in Sleep and Meditative States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Claassen, Associate Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RFA-AT-21-001
Record Dates: First submitted 2020-07-17; First posted 2020-08-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Sleep
Keywords: glymphatic system; meditation
MeSH Terms: conditions — Parkinson Disease | interventions — Meditation

STUDY DESIGN:
Masking Description: no masking is used in this protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adept Meditators (Experimental): Subjects will undergo scanning during awake, sleep deprived, and meditative states of consciousness.
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — meditation

SUMMARY:
This involves development and application of magnetic resonance imaging (MRI) methods for visualizing hemodynamic and metabolic relationships in healthy volunteers with advanced meditation experience.

DETAILED DESCRIPTION:
This study is evaluating the glymphatic system during awake, sleep, and meditative states.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-45
* "Adept meditator status"

Exclusion Criteria:

* Any non-MR compatible material implant, or contraindication to MR scanning
* Claustrophobia or inability to lie still for prolonged periods of time
* Participants with a recent (less than 2 months) infection, tattoo, or wound
* No consumption of stimulants or alcohol within 12 hours of the study visit
* clinical diagnosis of any major neurological or psychological condition
* Taking benzodiazepines, cholinestorase inhibitors, anti-psychotics, opioids, MAO inhibitors

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
CSF flow change | baseline to 24 hours
  Using MRI to assess the change in CSF flow in awake, sleep deprived, and meditative states

SECONDARY OUTCOMES:
EEG changes | baseline to 24 hours
  Looking at brain wave changes before and after intervention in Alpha, Beta, and Delta waves associated with light to deep sleep. The lowest bandwidth for alpha waves is 8 while the highest is 12. The lowest bandwidth for Beta waves is 13 Hz while the highest is 30 Hz. The lowest bandwidth for Delta waves is .4 Hz and the highest is 4 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Claassen, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No